CLINICAL TRIAL: NCT05801055
Title: Improvement in Endoscopic Mucosal Visibility Using a Pre-procedure Combination Drink of N-acetylcysteine and Simethicone: A Randomized Controlled Trial
Brief Title: A Study to Evaluate Endoscopic Visibility of Stomach After a Combination Drink of N-acetylcysteine and Simethicone
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2021-332-DM-124
Record Dates: First submitted 2023-03-06; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-02

CONDITIONS: Gastric Disease
Keywords: Endoscopy
MeSH Terms: conditions — Stomach Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Arm which will be randomised to get the combination drink prior to the diagnostic endoscopy
  Interventions: Drug: Evaluation of gastric visibility following the combination drink of N-acetyle cysteine and simethocone
- Arm 2 (No Intervention): Comparator arm where endoscopy will be done without any drink

INTERVENTIONS:
Drug: Evaluation of gastric visibility following the combination drink of N-acetyle cysteine and simethocone — The combination drink containing N-acetyl cysteine and simethicone help to disperse bubbles and mucus present in the stomach. During routine upper gastrointestinal endoscopy mucus and bubbles sometimes may hinder mucosal visibility, so small submucosal lesions, ulcers, erosions, and even flat pre-malignant lesions can be missed during endoscopy. The Japanese guidelines also recommend the use of this combination drink to detect early gastric cancers. So we plan to evaluate the role of this drink in improving gastric mucosal visibility in patients undergoing upper gastrointestinal endoscopy.
  Arms: Arm 1

SUMMARY:
Endoscopy is the diagnostic modality for most gastroduodenal diseases. During endoscopy mucus and foam may actually interfere with the visibility of the stomach mucosa. So the mixture of mucolytic ( N-acetyl cysteine) and anti-foaming agents ( simethicone) agents may disperse the bubbles and mucus in the stomach and enhance gastric visibility. This unique combination drink given 20-30 minutes prior to endoscopy is absolutely safe. There are previous studies from India, which was retrospective study. So, we have planned to conduct this randomized controlled trial on this issue. Adult patients undergoing diagnostic endoscopy will be randomized and one group (100 patients) will be given the combination drink whereas another group 9100 patients) will undergo an endoscopy after overnight fasting only, as a placebo drink may actually hamper the endoscopic visibility. Our primary outcome, gastric visibility will be assessed using a standard visibility scoring system.

DETAILED DESCRIPTION:
Improvement in endoscopic mucosal visibility using a pre-procedure combination drink of N-acetylcysteine and simethicone: A Randomized controlled trial

Introduction:

Upper gastrointestinal endoscopy (UGIE) is one of the most frequently performed procedures for diagnosing and treating GI and liver-related disorders. Pre-procedure preparation and reporting of adequate preparation is the standard of care for colonoscopies but there is not uniformity in preparation for UGIE. Various studies have demonstrated that the incidence of missed diagnosis in endoscopies can be brought down by improving mucosal visibility. Endoscopic mucosal visibility can be impaired by various factors like poor technique, excessive mucus, residual food, inappropriate positioning, and more importantly the presence of mucosal froth and bubbles in the GI tract. Gastro-duodenal mucosa is lined by mucus comprising 95% water and 5% cross-linked glycoprotein(GP), which keeps mucus viscous and liquid. With fasting, GP content decreases making mucus more sticky. Several mucolytic and anti-foaming agents including pronase, simethicone, and N acetyl-cysteine(NAC) have been tried for this purpose. NAC is a derivative of the natural amino acid L-cysteine. It breaks the disulfide bridges in high molecular weight glycoproteins. Simethicone (polydimethylsiloxane or dimethicone + SiO2) is an anti-foaming surface-acting agent, which acts by reducing the surface tension of air bubbles, surface viscosity, and hydrophobicity. Simethicone is virtually non-toxic, without any drug interaction or systemic toxicity. Multiple studies have been conducted showing the safety and efficacy of simethicone, NAC, and their combination for improving endoscopic visibility. These pre-medications are already used for improving endoscopic visibility to detect early esophageal and gastric cancer.

Some studies from the western countries as well as the eastern world have highlighted the significant role of mucolytic and anti-foaming agents in improving mucosal visibility.

Monrroy et al, in 2017 conducted a double-blind randomized control trial in which 230 patients were divided into 5 groups (46 each) i.e no intervention group, water 100 ml (W) group, and interventional groups comprised of simethicone alone (S), simethicone plus NAC 500 mg (S + NAC500) and simethicone plus NAC1000 group. The solution was ingested 20 minutes before the UGIE. Gastric visibility was assessed in 4 segments using a pre-validated mucosal visibility scoring system based on a Likert scale and adequate visibility was defined as a score less than 7. In this study, they found that premedication by S+NAC500 and S+NAC100 improved visibility whereas visibility was worst in the W group.

Another study by Manfredi et al in 2020 which was a prospective, endoscopist-blinded randomized study enrolled patients undergoing UGIE. Patients were randomized to receive NAC+S solution vs placebo. A pre-validated scoring system was used for the visibility assessment. A total score of less than 5 was considered insufficient preparation. The premeditated group had a significantly lower number of patients with a score <5. The need for water flush also occurred less in the premedicated group compared to the control group. One retrospective, investigator-blinded study was conducted in Sir Gangaram Hospital by Anikhindi et al in collaboration with Osaka International Cancer Institute, Osaka, Japan. It was designed as a case-control study. In this study group of patients who consumed 100 ml pre-endoscopy drink comprising of NAC + simethicone group were compared with the fasting group. Digital images were obtained from 6 pre-defined areas of the esophagus, stomach, and duodenum. A blinded investigator scored them using a 3-point scale for mucosal visibility. Mucosal visibility in the esophagus and stomach was significantly better in the NAC + S group compared to the 100 ml water group. There is no prospective data from India to validate the use of such pre-medications before routine UGIE. Therefore, we have designed a prospective randomized controlled trial to assess the improvement of mucosal visibility using a pre-endoscopic drink.

Need of the study:

Better visualization of the intestinal mucosa is important for diagnosing early changes of many benign lesions, precancerous lesions like Barrett's esophagus, or early flat malignant lesions. Most of the data about the role of NAC with simethicone are from Japan and the West, so studying this in the Indian population is required.

Aim of the study:

1. To clarify the role of NAC + S for better endoscopic mucosal visualization in the Indian population.

Study Methodology:

It will be a single-blind, parallel-randomized controlled trial. Randomization will be done using a table of random numbers. Using a computer-generated sequence. Allocation will be done through a sealed opaque envelope by a data entry operator to have allocation concealment (not the endoscopist or investigator).

The allocation ratio will be 1:1 between the study group and the control group. The study will be registered in a clinical trial registry after Institutional ethics clearance before the start of the study.

Study Centre: Department of Gastroenterology, Sanjay Gandhi Post Graduate Institute, Lucknow.

Duration of the study: May - June 2023 Sample size calculation The sample size has been calculated using OpenEpi Version 3 (CDC, Atlanta). The sample size was calculated taking the confidence limit (CL) of 99 %, power of the study of 95%, and alpha error of 5% to detect a 25% difference in adequate visibility between the study and control group, we got a minimum sample size of 174 (87 each group). Since we expect data loss and technical failure in 10-20% of patients we will include 100 patients in each group.

Inclusion criteria:

1. Consecutive patients presenting for ambulatory diagnostic endoscopy
2. Willing Informed consent
3. Age 18-75 years

Exclusion criteria:

1. Patients undergoing therapeutic endoscopy
2. Patients undergoing emergency endoscopy
3. Deeply sedated & anesthetized patients
4. Pregnant patients
5. Clinically suspected motility disorders (gastroparesis, achalasia)
6. Patients with esophageal stricture
7. Patients with gastric outlet obstruction.

Intervention: All patients will undergo a routine UGIE with the following instructions.

Upper GI endoscopy

* Overnight fasting
* Pharyngeal local anesthetic spray

Intervention Group:

Premedication with 15mL emulsions of NAC (600mg) + Simethicone (150 mg) diluted to 100 mL to be taken 10-30 mins prior to the procedure (not later).

Comparator:

The Control group will not receive any placebo emulsion as it has been shown to worsen the visibility.

Primary outcome:

The difference in adequate visibility between the two groups. Gastric total visibility score (TVS) 4-16 will be used as proposed by Monrroy et al [6]. The scoring system has been pre-validated to assess gastric endoscopic mucosal visibility. It will be calculated by assessment of mucosal visibility on a Likert scale of 1 to 4 in areas of the gastric antrum, lower gastric body, upper gastric body, and fundus (Figure 1).

It will be calculated by a blinded investigator using electronic images captured during the endoscopy.

A TVS <7 will be used to define adequate visibility (AV).

Secondary Outcome:

1. Time is taken for the procedure (scope-in-scope out)
2. Adverse events
3. Gastric mucosal lesion yield (%)

Statistical analysis All qualitative data will be presented as proportions and quantitative data will be expressed as mean (± standard deviation) or median (interquartile range) as appropriate. Adequate visibility, gastric lesion yield, and adverse events between the group will be compared using the Chi-squared test. The time taken for the procedure between the two groups will be compared using the Mann-Whitney U test. A power of 80% and an alpha error of 5% is permitted. A p-value of <0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive patients presenting for ambulatory diagnostic endoscopy
2. Willing Informed consent
3. Age 18-75 years

Exclusion Criteria:

1. Patients undergoing therapeutic endoscopy
2. Patients undergoing emergency endoscopy
3. Deeply sedated & anesthetized patients
4. Pregnant patients
5. Clinically suspected motility disorders (gastroparesis, achalasia)
6. Patients with esophageal stricture
7. Patients with gastric outlet obstruction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Any change in adequate visibility between the two groups. | Upto three months
  The difference in adequate visibility between the two groups. Gastric total visibility score (TVS) will be used as proposed by Monrroy et al. It will be calculated by assessment of mucosal visibility on a Likert scale of 1 to 4 in areas of the gastric antrum, lower gastric body, upper gastric body and fundus. A TVS <7 will be used to define adequate visibility (AV).

SECONDARY OUTCOMES:
Any change in endoscopy time | Upto one week
  1.Time taken for the procedure (scope-in-scope out)
The rate of adverse outcome | Upto one week
  To look for any adverse outcomes and compare between two group
The rate of gastric mucosal lesion yield | Upto one week
  We will also compare if gastric mucosal lesion yield is different in the interventional arm compared to the '' no drink'' group

CONTACTS AND LOCATIONS:
Locations (1):
- Sanjay Gandhi Postgraduate Institute of Medical Sciences (SGPGIMS), Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monrroy H, Vargas JI, Glasinovic E, Candia R, Azua E, Galvez C, Rojas C, Cabrera N, Vidaurre J, Alvarez N, Gonzalez J, Espino A, Gonzalez R, Parra-Blanco A. Use of N-acetylcysteine plus simethicone to improve mucosal visibility during upper GI endoscopy: a double-blind, randomized controlled trial. Gastrointest Endosc. 2018 Apr;87(4):986-993. doi: 10.1016/j.gie.2017.10.005. Epub 2017 Oct 14. PMID 29037773
- [Result] Anikhindi SA, Kumar A, Uedo N, Singla V, Anikhindi A, Sharma P et al. Pre-endoscopy drink of simethicone and N-acetylcysteine significantly improves visualization in upper gastrointestinal endoscopy. J Dig Endosc. 2021;12(1):11-8. doi: 10.1055/s-0041-1726225.